CLINICAL TRIAL: NCT03280784
Title: Clinical Audit on the Use of Upper Gastrointestinal Endoscopy in Assiut University Children Hospital
Brief Title: Clinical Audit on the Use of Upper Endoscopy in Assist University Children Hospital
Acronym: CAOUOEUIAUCH
Status: Completed | Type: Observational
Sponsor: Mahmoud Mohammed Osman Ali (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Mohammed Osman Ali, principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU Pediatric hospital
Record Dates: First submitted 2017-09-07; First posted 2017-09-13 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Upper Gastrointestinal Endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this protocol aides to evaluate:( 1)whether upper gastrointestinal endoscopy (UGE) is used appropriately according to the Guideline on pediatric GI endoscopy [1] commissioned by the European Society for Paediatric Gastroenterology Hepatology and Nutrition(ESPGHAN) and the European Society of Gastrointestinal Endoscopy(ESGE). In our hospital setting and(2) whether there is any relationship between appropriateness of gastrointestinal endoscopy and the presence of lesions detected by endoscopy.

DETAILED DESCRIPTION:
gastrointestinal endoscopy is a safe and effective procedure. However,complications do exist and procedure-related costs are significant The rapid escalation of the cost of medical care, in the face of limited resources, is making the appropriateness of indications more and more essential to the rational utilization of such resources.Upper Gastrointestinal (UGI) endoscopy in the pediatric population has evolved during the last 30 years with an increasing number of diagnostic and therapeutic applications.

years with an increasing number of diagnostic and therapeutic Technological improvements and endoscopic devices have contributed to the evolution This prospective study is to determine whether upper gastrointestinal endoscopy is used appropriately in our hospital setting according to, the Guideline on pediatric GI endoscopy [1] commissioned by the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) and the European Society of Gastrointestinal Endoscopy (ESGE). and whether the appropriateness of use Predicts the probability of detecting significant lesions by endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Weight loss,

failure to thrive

Unexplained anemia

Abdominal pain with suspicion of an organic disease

Dysphagia or odynophagia

Caustic ingestion

Recurrent vomiting exclusion criteria

patients with perforated viscous

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children admitted at assiut university hospital for upper gastrointestinal endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
improve the use of upper gastrointestinal endoscopy in assiut university hospital of upper gastrointestinal endoscopy in assiut university children hospital | One year
  appropriateness
  This prospective study is to determine whether upper gastrointestinal endoscopy is used appropriately in our hospital setting according to, the Guideline on pediatric GI endoscopy [1] commissioned by the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) and the European Society of Gastrointestinal Endoscopy (ESGE). and whether the appropriateness of use Predicts the probability of detecting significant lesions by endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud mohammed, MD, Principal Investigator — Assiut
Locations (1):
- Assiut university children hospital, Asyut, Egypt